CLINICAL TRIAL: NCT01353690
Title: A Prospective, Multicenter, Feasibility Study of Autologous Muscle-derived Cell (AMDC) Transplantation for Treatment of Advanced Ischemic Heart Failure
Brief Title: Autologous Cell Therapy for Ischemic Heart Failure
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cook MyoSite (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-013
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Ischemic Heart Disease
Keywords: Cell Therapy; Heart Failure; Heart Disease; Myocardial Infarction; Myocardial Ischemia; Autologous; Muscle-derived Cell
MeSH Terms: conditions — Myocardial Ischemia; Heart Failure; Heart Diseases; Myocardial Infarction

ARMS (1):
- AMDC (Experimental)
  Interventions: Biological: AMDC

INTERVENTIONS:
Biological: AMDC — Cell Treatment

SUMMARY:
The aim of this clinical study is to investigate the safety and feasibility of Autologous Muscle-derived Cells (AMDC; a preparation of a patient's own cells) as a treatment for patients with advanced heart failure caused by ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 but less than 80 years
* Prior myocardial infarction
* Depressed left ventricular ejection fraction (LVEF) ≤ 35%
* NYHA functional classification of II to IV

Exclusion Criteria:

* Not under stable optimal medical management
* Cardiac surgery or percutaneous coronary intervention within 3 months
* Occurrence of myocardial infarction (MI) within 6 months, in the case of first MI, or 3 months, in the case of any subsequent MI
* Prior cell, gene, or transmyocardial laser revascularization therapy
* Ventricular wall thickness in target region ≤ 5 mm
* Moderate to severe aortic valve stenosis or mechanical valve replacement
* Left ventricular aneurysm or thrombus
* Left ventricular dysfunction associated with a reversible cause
* Vascular disease preventing percutaneous vascular access
* History of myopathic disease
* History of neoplasia within 5 years, except for basal cell carcinoma
* Receiving or planning to receive anti-cancer medications
* Serum creatinine > 3.0 mg/dl
* Pregnant, planning to become pregnant, or breastfeeding a child in the next 18 months
* Life expectancy of less than 1 year
* Morbid obesity (defined as BMI > 35)
* History of bleeding diathesis or coagulopathy
* Positive for HIV, Hepatitis B, or Hepatitis C
* Known hypersensitivity or contraindication to study product or treatment procedure
* Enrolled in another research project at the time of enrollment
* Unable to provide informed consent
* Unable or unwilling to commit to the follow-up clinical procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-02-05 (Actual); Primary Completion 2012-12-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Incidence of major adverse events associated with the use of AMDC | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Hung Q. Ly, MD, Principal Investigator — Montreal Heart Institute
Locations (2):
- Canada (2):
  - University of Alberta and Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - Montreal Heart Institute, Montreal, Quebec